CLINICAL TRIAL: NCT05841615
Title: Evaluation of the Safety and Efficacy of Pulmonary Vein Isolation (PVI) Combined With Renal Denervation (RDN) in Patients With Atrial Fibrillation (AF) and Hypertension (HTN)
Brief Title: Pulmonary Vein Isolation (PVI) Combined With Renal Denervation (RDN) in Atrial Fibrillation (AF) and Hypertension (HTN)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Zhengrong Huang, Professor, The First Affiliated Hospital of Xiamen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-RDN and PVI
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: AF - Atrial Fibrillation; HTN-Hypertension
Keywords: Pulmonary Vein Isolation (PVI); Renal Denervation (RDN); Atrial Fibrillation (AF); Hypertension (HTN)
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI alone (Sham Comparator): Participants only experience PVI operations
  Interventions: Other: Pulmonary vein isolation
- PVI and RDN (Experimental): Participants experience both PVI and RDN operations
  Interventions: Other: Renal Denervation operation; Other: Pulmonary vein isolation

INTERVENTIONS:
Other: Renal Denervation operation — RDN: Percutaneous renal artery sympathetic radiofrequency ablation for both sides. For each side, a total of 13 targets were ablated. The ablation power was 8W~12W for 40 seconds
  Arms: PVI and RDN
Other: Pulmonary vein isolation — PVI: Pulmonary vein isolation was performed until the potential of each pulmonary vein disappeared under the guidance of the CARTO mapping system. Ablation of the top line and the bottom line of the left atrium was performed at the same time.

SUMMARY:
The close relationship between the increase of sympathetic tension, AF, and HTN cannot be ignored. In addition, the significant failure rate of PVI (20-50%) in the treatment of AF makes it very necessary to explore the effect of RDN on AF. Therefore, this study aims to compare the effects and safety of PVI alone and PVI combined with RDN with AF combined with HTN, which will open a new chapter for PVI combined with RDN in the treatment of AF.

ELIGIBILITY:
Inclusion Criteria:

* 18<age<75years
* clinic blood pressure≥140/90mmHg or 24-hour ambulatory blood pressure monitoring average blood pressure ≥135/85mmHg
* Ecg diagnosis of atrial fibrillation ;
* who signed informed consent and were approved by the Ethics Committee of the First Affiliated Hospital of Xiamen University.

Exclusion Criteria:

* pregnant women or lactating patients;
* Patients who were unsuitable for ablation before surgery （unilateral or bilateral renal artery shape and structure were found： renal artery stenosis exceeding 50%, renal aneurysm, previous renal artery interventional surgery, renal artery malformation, renal artery diameter < 4mm or length of treatable segment < 20mm）
* Patients who only have one kidney or have a history of kidney transplantation
* Patients with a history of renal arterial intervention or renal denervation
* identified secondary hypertension or Pseudo hypertension except for renal parenchymal hypertension;
* malignant tumors or end-stage diseases;
* Severe peripheral vascular disease, abdominal aortic aneurysm
* whose left atrium is larger than 55mm
* obvious bleeding tendency and blood system diseases;
* Severe peripheral vascular disease, abdominal aortic aneurysm;
* A history of the acute coronary syndrome within two weeks;
* acute or severe systemic infection;
* drug or alcohol dependence or refusal to sign informed consent.
* Other conditions that are not suitable for PVI and RDN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Malignant end point event 1 | within 2 years post operation
  Fatal and nonfatal stroke
Malignant end point event 2 | within 2 years post operation
  cerebral hemorrhage
Malignant end point event 3 | within 2 years post operation
  acute myocardial infarction
Malignant end point event 4 | within 2 years post operation
  cardiovascular death

SECONDARY OUTCOMES:
Complex end point event 1 | within 2 years post operation
  Hospitalization for heart failure
Complex end point event 2 | within 2 years post operation
  elevation of blood pressure(mmHg, upper arm blood pressure electronic monitor)
Complex end point event 3 | within 2 years post operation
  left ventricular hypertrophy(mm, by Cardiac color ultrasound)
Complex end point event 4 | within 2 years post operation
  coronary revascularization(by coronary arteriography)
Complex end point event 5 | within 2 years post operation
  transient ischemic attack
Complex end point event 6 | within 2 years post operation
  renal insufficiency (eGFR ml/min, by ECT);
Complex end point event 7 | within 2 years post operation
  renal artery stenosis(by renal arteriography)
Complex end point event 8 | within 2 years post operation
  proteinuria(mg/L, PRM assay)
Complex end point event 9 | within 2 years post operation
  the recurrence rate of atrial fibrillation
Complex end point event 10 | within 2 years post operation
  the control rate of blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hopital of Xiamen University, Xiamen, Fujian, China